CLINICAL TRIAL: NCT06073977
Title: Risk Factors for Pediatric Difficult Supraglottic Airway Placement and Ventilation (PEDSGAP): A Multicentric Prospective Observational Study
Brief Title: Risk Factors for Pediatric Difficult Supraglottic Airway Placement and Ventilation
Acronym: PEDSGAP
Status: Completed | Type: Observational
Sponsor: Alper Kilicaslan (Other)
Collaborators: Emre Sertaç Bingül (Unknown); Nüzhet Mert Şentürk (Unknown); Sibel Seçkin Pehlivan (Unknown); Şengül Özmert (Unknown); Özlem Sezen (Unknown); Gaye Aydın (Unknown); Esra Turunç (Unknown); Faruk Çiçekçi (Unknown); Sedat Saylan (Unknown); Alkin Çolak (Unknown)
Responsible Party: Sponsor-Investigator, Alper Kilicaslan, Prof, Konya Necmettin Erbakan Üniversitesi
Organization: Konya Necmettin Erbakan Üniversitesi (Other)
Other Study IDs: 2023/4546
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Laryngeal Mask Airway; Children; Airway Management
Keywords: Supraglottic Airway; Laryngeal Mask Airway; Children; Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to observe the occurrence of failure or difficulty during placement of supraglottic airway devices (SGAs) and its associated risk factors in pediatric patients. Despite wide use in pediatric practice, not much is known related to problems during SGA insertion unlike adults. The main information regarding pediatric SGA comes from either small comparative studies or retrospective studies reporting increased risk of failure. Thus the main aim of this prospective, multicentric, observational study is to determine the incidence of "difficult" or "failed" SGA placement in children and clarify the possible risk factors for difficulty.

DETAILED DESCRIPTION:
Inclusion criteria

* 1- 12 years old peditatric patients
* ASA class I- III
* Scheduled for elective surgery under general anaesthesia, in whom a SGA would be used for airway maintenance
* Planned surgery under general anesthesia with SGA
* Patients whose legal guardians provide informed consent

Exclusion criteria

* Refusal to participate in the study.
* Inability of patient or parents to understand the study or consent process
* Orotracheal intubation requirement
* Pathology of airway, neck, respiratory tract, upper gastrointestinal tract
* Increased risk of regurgitation or aspiration
* Emergency surgeries
* Requirement for intensive care follow-up after the surgery

ELIGIBILITY:
Inclusion Criteria:

* 1- 12 years old peditatric patients
* ASA class I- III
* Planned surgery under general anesthesia with supraglottic airway
* Patients whose legal guardians provide informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Inability of patient or parents to understand the study or consent process
* Orotracheal intubation requirement
* Pathology of airway, neck, respiratory tract, upper gastrointestinal tract
* Increased risk of regurgitation or aspiration

  * Emergency surgeries
  * Requirement for intensive care follow-up after the surgery

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1- 12 years old peditatric patients scheduled for elective surgery under general anaesthesia, in whom a SGA would be used for airway maintenance
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The incidence of difficulty in supraglottic airway device(SGA) placement | Immediately after the attempt of insertion and up to the end of the surgery
  Difficulty in placing SGA is defined as follows: SGA insertion that requires more than one attempt,need for a change the size or type of SGA,desatutaion (SpO2<93%), disrupted capnography,high airway pressure (>25 cmH2O of peak pressure)

SECONDARY OUTCOMES:
Risk factors for pediatric difficult SGA placement | At the beginning of anesthesia
  Possible risk factors related with failure and difficulty listed as:experience of the anaesthetist , presence of history of asthma/pneumoniae,presence of craniofascial anomalies, use of neuromuscular blocking agent, type and placement technique of SGA
The incidence of complications related to SGA insertion | Up to 24 hours after surgery
  The incidence of adverse events including laryngospasm, desaturation bronchospasm, stridor, regurgitation bucking, airway trauma and postoperative complications including difficult weaning, cough, stridor, vomiting, dysfagia, dysphonia

CONTACTS AND LOCATIONS:
Overall Officials: Alper Kilicaslan, Principal Investigator — Necmettin Erbakan Universty Medical Faculty
Locations (6):
- Turkey (Türkiye) (6):
  - Asli Dönmez, Ankara
  - Emre Sertaç Bingül, Istanbul
  - Gaye Aydin, Izmir
  - Sibel Seçkin Pehlivan, Kayseri
  - Necmettin Erbakan University, Konya
  - Sedat Saylan, Trabzon